CLINICAL TRIAL: NCT05306327
Title: Neurologic Physiology After Removal of Therapy (NeuPaRT): Pilot Multicentre Feasibility Study
Brief Title: Neurologic Physiology After Removal of Therapy (NeuPaRT)
Acronym: NeuPaRT
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: Reda 12243
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Determination of Death
MeSH Terms: conditions — Death | interventions — Electroencephalography; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: electroencephalography (EEG) — 1. brain cortical activity using full scalp
  2. cerebral blood flow velocity
  3. during the dying process following planned withdrawal of life sustaining measures (WLSM)
  Other Names: transcranial Doppler (TCD); related (EP), somatosensory (SSEP)

SUMMARY:
The purpose of this study is to determine when brain function stops compared to when the heart stops by monitoring electrical brain activity in patients who are taken off life support and progress to death in the intensive care unit.

DETAILED DESCRIPTION:
There are many Canadians who need an organ transplant and who will never get one. In the past, people could only be organ donors after being declared brain dead.

The dead donor rule serves this purpose by ensuring that death determination precedes organ retrieval. In Canada, death determination occurs in one of two ways. In neurologic determination of death (NDD), death is declared upon completion of a standardized neurologic assessment that confirms permanent loss of brain activity. In donation after circulatory determination of death (DCDD), death is declared 5 minutes after circulatory arrest. By confirming permanent loss of brain activity, the current NDD process protects donors from suffering and maintains stakeholder trust. In contrast, the current DCDD process assumes, but does not explicitly confirm, permanent loss of brain activity when death is declared 5 minutes after circulatory arrest. While this assumption is rooted in a strong physiologic rationale, lack of compelling evidence regarding cessation of brain activity in humans contributes to ongoing mistrust of the DCDD process among healthcare and public stakeholders.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Plan for the withdrawal of life sustaining measures (WLSM)
3. Attending physician anticipates patient will die within 24 hours of the withdrawal of life sustaining measures
4. Patient has an indwelling arterial cannula for monitoring blood pressure

Exclusion Criteria:

1. Brain death or plan for Neurologic Determination of Death (NDD)
2. Injuries that anatomically preclude the use of neurologic monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients admitted to a participating ICU who fulfil all the inclusion criteria and for whom none of the exclusion criteria exist.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Patient Accrual complete study procedures) | 2022 to 2023
  90 patients at all sites and an additional 18 patients at the lead site for specific tests

SECONDARY OUTCOMES:
Waveform Data Completeness | 2022-2023
  Adequate waveform signal that (i) spans circulatory arrest, (ii) includes data for at least 80% of the planned observation period (from the withdrawal of life sustaining measures to 30 minutes after circulatory arrest [or 5 minutes for confirmed donation after circulatory determination of death (DCDD) donors]), and (iii) has a clearly identifiable time of cessation for each signal.
Time Difference Circulatory Arrest and Cessation of EEG Activity | 2022-2023
  Cerebral blood flow velocity in middle cerebral artery (when available), and cessation of event/evoked potentials (LHSC site only). See below for definition of cessation of each signal.

CONTACTS AND LOCATIONS:
Overall Officials: Teneille Gofton, MD MSc FRCPC, Principal Investigator — London Health Sciences Centre
Locations (5):
- Canada (5):
  - University of Calgary Foothills Campus, Calgary, Alberta
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Centre hospitalier de l'Université de Montréal,, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing should be directed to the principal investigator (Dr. T. Gofton) and will be considered on a case by case basis and with approval from the Western Health Sciences Research Ethics Board. No video will be shared at any time.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of data analysis (5 years after study initiation August 2022)

REFERENCES:
- [Derived] Gofton T, Dhanani S, Meade M, Boyd JG, Chamberlain E, Chandler J, Chasse M, Scales NB, Choi YH, D'Aragon F, Debicki D, English S, Fantaneanu TA, Kramer AH, Kromm J, Murphy N, Norton L, Singh J, Smith MJ, Weijer C, Shemie S, Bentall TC, Campbell E, Slessarev M. Neurologic Physiology after Removal of Therapy (NeuPaRT) study: study protocol of a multicentre, prospective, observational, pilot feasibility study of neurophysiology after withdrawal of life-sustaining measures. BMJ Open. 2023 Apr 27;13(4):e073643. doi: 10.1136/bmjopen-2023-073643. PMID 37105694